CLINICAL TRIAL: NCT03284944
Title: Small-Volume Tubes to Reduce Anemia and Transfusion (STRATUS): A Pilot Study
Brief Title: Small-Volume Tubes to Reduce Anemia and Transfusion (STRATUS)
Status: Completed | Type: Observational
Sponsor: Population Health Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: STRATUS Pilot
Record Dates: First submitted 2017-07-09; First posted 2017-09-15 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Blood Loss Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control (Before) Period: Use of standard-volume blood collection tubes (6 weeks)
  Interventions: Device: Standard-Volume
- Intervention (After) Period: Use of small-volume ("soft-draw") blood collection tubes (6 weeks following 2-week washout period)
  Interventions: Device: Small-Volume

INTERVENTIONS:
Device: Small-Volume — Small-volume (2 - 3 mL "soft-draw" Vacutainer tubes, Beckton Dickinson) ethylenediaminetetraacetic acid (EDTA), lithium-heparin, citrate, fluoride and silica tubes.
  Groups: Intervention (After) Period
Device: Standard-Volume — Standard-volume (4 - 6 mL Vacutainer tubes, Beckton Dickinson) ethylenediaminetetraacetic acid (EDTA), lithium-heparin, citrate, fluoride and silica tubes.
  Groups: Control (Before) Period

SUMMARY:
STRATUS will evaluate the use of small-volume ("soft-draw") blood collection tubes for laboratory testing in reducing anemia and transfusion in intensive care unit patients without significant adverse consequences. This is a simple, cost-neutral intervention that could improve the quality of patient care and reduce the harms of frequent laboratory testing.

DETAILED DESCRIPTION:
The STRATUS Pilot Study is a prospective observational study (before-after design) to assess the feasibility of implementing a full-scale randomized trial powered for clinical outcomes (RBC transfusion, incidence and severity of anemia). Identification of barriers and facilitators of implementation will enhance the conduct of the full-scale trial and facilitate incorporation of the intervention into routine practice.

ELIGIBILITY:
Investigative Site Eligibility:

* Intensive care unit with at least 15 beds with capacity for mechanical ventilation
* Current standard to use standard-draw blood collection tubes
* Availability of hospital administrative data and electronic patient information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients admitted to the participating intensive care unit at the investigative site.
Sampling Method: Non-Probability Sample
Enrollment: 369 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-02-07 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Successful crossover from standard-volume to small-volume tubes | 2 week washout period
  Defined as at least 95% correct tubes collected during an audit of tubes in the storage area at the end of the washout period
Adherence to the correct tube size during the intervention period | 6 week intervention period
  Defined as at least 95% adherence to allocated tube size evaluated during audits of tubes in the storage area
Sufficient volume for testing with small-volume tubes | 6 week intervention period
  Defined as <3% of samples reported as inadequate volume for testing
Acceptability of the intervention by end-users | 6 week intervention period
  Acceptability qualitatively evaluated during structured focus group discussions
Complete primary data collection | 14 weeks
  Defined as at least 95% of patients with complete data collected

SECONDARY OUTCOMES:
Reduction in blood loss | 12 weeks
  Reduction in blood loss from routine hematology, chemistry, and coagulation testing using small-volume tubes.
RBC units transfused | 12 weeks
  Number of RBC units transfused per patient-day in the ICU.
Change in hemoglobin | 12 weeks
  Change in hemoglobin level from ICU admission to ICU discharge (or death) adjusted for RBC transfusion.
ICU and hospital length of stay | 12 weeks
  ICU and hospital length of stay
ICU and hospital mortality | 12 weeks
  ICU and in-hospital mortality

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Siegal, MD, Principal Investigator — Population Health Research Institute, McMaster University, Hamilton Health Sciences; Stuart Connolly, MD, Principal Investigator — Population Health Research Institute, McMaster University, Hamilton Health Sciences
Locations (1):
- Hamilton Health Sciences - Hamilton General Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Siegal DM, Belley-Cote EP, Lee SF, Robertson T, Hill S, Benoit P, Meeks B, Owen J, Roglich T, Zotova E, Connolly SJ. Small-volume tubes to reduce anemia and transfusion (STRATUS): a pilot study. Can J Anaesth. 2023 Nov;70(11):1797-1806. doi: 10.1007/s12630-023-02548-6. Epub 2023 Jul 28. PMID 37505420